CLINICAL TRIAL: NCT03915561
Title: Effect of Intravenous Dynastat on Postoperative Sore Throat: A Randomized Double-blinded Controlled Trial
Brief Title: Effect of Intravenous Dynastat on Postoperative Sore Throat
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Po-Kai Wang, Head of Pain Management, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB108-27-A
Record Dates: First submitted 2019-03-31; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Sore Throat; Postoperative Complications
Keywords: postoperative sore throat
MeSH Terms: conditions — Pharyngitis; Postoperative Complications | interventions — parecoxib; Saline Solution

STUDY DESIGN:
Intervention Model Description: a two-arm, individually randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list will be generated using computer sequence number, and patient allocation ratio will be 1:1. Written allocation group will be sealed in individual opaque envelopes marked externally only with study identification numbers. An anesthetic assistant not participating in the study prepared the drug solution after breaking the codes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): This group will be received intravenous injection with 10ml transparent mixture solution with 40mg Dynastat and 0.9% saline twice
  Interventions: Drug: Parecoxib Injectable Product
- Placebo (Placebo Comparator): This group will be received intravenous injection with 10ml 0.9% saline alone (transparent solution) twice
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Parecoxib Injectable Product — Dynastat (parecoxib sodium) is rapidly converted to valdecoxib following injection and reduces the production of prostaglandins that are important mediators of pain and inflammation. After intravenous injection with 40mg Dynastat, the onset of analgesia was 7-14 minutes and reached a peak effect within 2 hours. After a single dose, the duration of analgesia was dose and clinical pain model dependent and ranged from 6 to greater than 24 hours and maximal daily dose of Dynastat is 80mg. According to recommendation of acute postoperative pain management and product information, the timing of first injection will be at 10 minutes before anesthetic induction, and second injection will be 6 to 12 hours after first injection.
  Other Names: Dynastat
  Arms: Study group
Drug: Normal saline — Placebo group (0.9% saline, group S) will be received intravenous injection with 10ml 0.9% saline alone (transparent solution) twice.
  Arms: Placebo

SUMMARY:
A postoperative sore throat (POST) after tracheal intubation is one of the most common postoperative problems causing dissatisfaction to participants, including sore throat, dry throat, cough, sputum, hoarseness and even dysphagia. Both nonpharmacological and pharmacological measures have been attempted to alleviate the incidence and severity of POST with variable success. Airway inflammation may be important in the pathogenesis of these symptoms in intubated participants but however, there was still no study to investigate the effect of cyclooxygenase-2 (COX-2) for the prevention of POST. So, the investigators' study will be the first one to investigate if perioperatively intravenous (IV) Dynastat injection can be used as a new indication for POST prevention.

DETAILED DESCRIPTION:
The investigators' study will be designed a two-arm, individually randomized, double-blind, placebo-controlled trial comparing two doses of 40mg Dynastat with placebo (0.9% saline) in participants who will receive noncardiac surgery under general anesthesia with tracheal intubation. The investigators will include participants of American Society of Anesthesiologists physical status 1 and 2, 20-65 years of age, requiring general anesthesia with endotracheal intubation (ETGA) for elective non-cardiac surgery will be enrolled. Besides, the anesthetic time after intubation will need 90 minutes at least. Those with a preexisting cough, hoarseness or a sore throat, smoker, history of asthma or chronic obstructive pulmonary disorder, vocal performer by occupation, recent or recurrent respiratory tract infection, risk factors for postoperative aspiration, obesity, pregnancy, and contraindication to Dynastat medications will be excluded. Anticipated difficult intubation, Mallampati grade >2, difficult mask ventilation requiring oral or nasal airway, Cormack and Lehane grade III and IV on laryngoscopy, intubation attempt >1, moderate to severe liver dysfunction (Child-Pugh score >7), severe renal dysfunction (Ccr < 30 ml/min), congestive heart failure (NYHA II-IV), and those requiring orogastric or nasogastric tubes will be other exclusion criteria. In the operating room, participants will receive study drug according to the group allocation. General anesthesia will be induced with IV fentanyl 2 μg/kg and propofol 2 mg/kg, followed by rocuronium 0.8 mg/kg. After achieving adequate time of neuromuscular blockade onset, an anesthesiologist (endotracheal tube intubation numbers > 500 times), unaware of the group allocation, will perform laryngoscopy in all the groups using standard 3 or 4 Macintosh blades. Polyvinylchloride endotracheal tubes (ETTs) with a 7-mm ID for male and 6.5-mm ID for female will be used for orotracheal intubation. Lubrication will be applied on the ETT. The cuff will be inflated with air to the point just capable of sealing leakage. The cuff pressure will be checked and adjusted to 25-30 cmH2O with the help of pressure gauge. At the end of surgery, the residual neuromuscular block will be antagonized with IV neostigmine 0.05 mg/kg and glycopyrrolate 0.01 mg/kg. Gentle suctioning of oral secretions will be done with 12F soft suction catheter while limiting the suction pressure to 50 cmH2O before tracheal extubation. After tracheal extubation, participants will be transferred to the postanesthetic care unit. The following variables at the time of tracheal intubation and extubation will be recorded: Cormack and Lehane laryngoscopy score; resistance to ETT insertion (none/mild/moderate); the time to achieve intubation will be defined as the time from opening of mouth for insertion of laryngoscope blade to confirmed placement of ETT (assessed with chest auscultation and capnograph); application of external laryngeal pressure to aid endotracheal intubation; duration of tracheal intubation defined as the time from placement of ETT to its removal; repositioning of ETT; blood tinge on the suction catheter during oral suctioning; blood stain on ET after its removal; and total opioid consumption in the postoperative period. The investigators' primary subject will be the incidence of POST, and the main effects of Dynastat will be the primary interest. The incidence of POST will be also compared among the 2 groups. Secondary outcomes included the severity of POST, incidences and severity of cough, hoarseness, and dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 and 2
* Requiring general anesthesia with endotracheal intubation (ETGA) for elective non-cardiac surgery
* The anesthetic time after intubation will need 90 minutes at least.

Exclusion Criteria:

* Those with a preexisting cough, hoarseness or a sore throat
* Smoker
* History of asthma or chronic obstructive pulmonary disorder
* Vocal performer by occupation
* Recent or recurrent respiratory tract infection
* Risk factors for postoperative aspiration, for example obesity, pregnancy
* Allergic reaction to Dynastat, acetylsalicylic acid, sulfonamide or NSAIDs.
* Active GI bleeding or gastric ulcer
* Third trimester and during lactation
* Anticipated difficult intubation
* Mallampati grade >2
* Difficult mask ventilation requiring oral or nasal airway
* Cormack and Lehane grade III and IV on laryngoscopy
* Intubation attempt >1
* Moderate to severe liver dysfunction (Child-Pugh score >7)
* Severe renal dysfunction (Ccr < 30 ml/min)
* Congestive heart failure (NYHA II-IV)
* Those requiring orogastric or nasogastric tubes

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
The early incidence of POST | The early incidence will be assessed between 1 and 2 hours after surgery
  The early incidence of POST will be also compared among the 2 groups
The late incidence of POST | The late incidence will be assessed at 24 hours after surgery
  The late incidence of POST will be also compared among the 2 groups

SECONDARY OUTCOMES:
The early severity of POST | The early severity of POST will be assessed between 1 and 2 hours after surgery
  0 to 100, 0 = no POST at any time since the operation, and 100 = the most severe POST after the operation
The late severity of POST | The late severity will be assessed at 24 hours after surgery
  0 to 100, 0 = no POST at any time since the operation, and 100 = the most severe POST after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Po-Kai Wang, PhD, Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Po-Kai Wang, Hualien City, Hualien, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tanaka Y, Nakayama T, Nishimori M, Tsujimura Y, Kawaguchi M, Sato Y. Lidocaine for preventing postoperative sore throat. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD004081. doi: 10.1002/14651858.CD004081.pub3. PMID 26171894
- [Result] Hara K, Maruyama K. Effect of additives in lidocaine spray on postoperative sore throat, hoarseness and dysphagia after total intravenous anaesthesia. Acta Anaesthesiol Scand. 2005 Apr;49(4):463-7. doi: 10.1111/j.1399-6576.2005.00632.x. PMID 15777293
- [Result] McHardy FE, Chung F. Postoperative sore throat: cause, prevention and treatment. Anaesthesia. 1999 May;54(5):444-53. doi: 10.1046/j.1365-2044.1999.00780.x. PMID 10995141
- [Result] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989
- [Result] Cheer SM, Goa KL. Parecoxib (parecoxib sodium). Drugs. 2001;61(8):1133-41; discussion 1142-3. doi: 10.2165/00003495-200161080-00010. PMID 11465874
- [Result] Harris SI, Stoltz RR, LeComte D, Hubbard RC. Parecoxib sodium demonstrates gastrointestinal safety comparable to placebo in healthy subjects. J Clin Gastroenterol. 2004 Aug;38(7):575-80. doi: 10.1097/00004836-200408000-00007. PMID 15232360
- [Result] Graff J, Arabmotlagh M, Cheung R, Geisslinger G, Harder S. Effects of parecoxib and dipyrone on platelet aggregation in patients undergoing meniscectomy: a double-blind, randomized, parallel-group study. Clin Ther. 2007 Mar;29(3):438-47. doi: 10.1016/s0149-2918(07)80082-8. PMID 17577465
- [Result] Schug SA, Joshi GP, Camu F, Pan S, Cheung R. Cardiovascular safety of the cyclooxygenase-2 selective inhibitors parecoxib and valdecoxib in the postoperative setting: an analysis of integrated data. Anesth Analg. 2009 Jan;108(1):299-307. doi: 10.1213/ane.0b013e31818ca3ac. PMID 19095866